CLINICAL TRIAL: NCT04928404
Title: Barbed Suspension of the Tongue Base for Treatment of Obstructive Sleep Apnea Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abd Elmateen Moussa, Otorhinolaryngology specialist, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-med-21-06-12
Record Dates: First submitted 2021-06-15; First posted 2021-06-16 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: tongue base; tongue base suspension; barbed suture
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obstructive sleep apnea patients (Other)
  Interventions: Procedure: tongue base suspension using barbed suture

INTERVENTIONS:
Procedure: tongue base suspension using barbed suture — all patients will undergo multi-level surgeries .Therefor, Anterolateral advancement pharyngeoplasty (ALA) or Barbed Reposition Pharyngoplasty (BRP) will be applied to improve retro-palatal obstruction and tongue base suspension using barbed suture for retro-lingual obstruction.

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common clinical condition in which the throat narrows or collapses repeatedly during sleep, causing obstructive sleep apnea events.

One of the most common sites for collapse during sleep is hypo-pharyngeal space. It was founded in 50% of OSA patients those have moderate and severe apnea.

DeRowe et al invented the Tongue base suspension operation in 1998 for sleep disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* BMI of patients less than 35 kg/m2.
* Patients who have symptoms and signs of OSA.
* Moderate to severe OSAHS confirmed by formal polysomnography (defined as an AHI ≥15).
* Friedman tongue position III or IV.
* Documented failure/refusal of attempts of conservative treatment measures (not limited to continuous positive airway pressure).
* The presence of retrolingual collapse confirmed preoperatively with flexible fiberoptic endoscope during Muller maneuver.
* Patients have macroglossia as defined by posterior airspace (PAS) of ≤10mm.

Exclusion Criteria:

* Failure to attend postoperative follow-up polysomnography within 6 months of surgery.
* Previous surgery to the base of the tongue or other surgical treatment of OSAHS.
* A history of malignancy or infection of the head and neck region, laryngeal trauma, or other previous oropharyngeal/laryngeal surgery.
* Patients have retrognanthia sella-nasion-supra mentale (SNB) ≥76º.
* Huge lymphoid tissue of the tongue and/or lingual tonsil.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
changes in obstructive sleep apnea | 3 months after intervention
  using polysomnography

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol